CLINICAL TRIAL: NCT01275833
Title: Restoration of Atrioventricular Synchrony Trial
Acronym: RESTORE-AV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult subject recruitment
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: RESTORE AV
Record Dates: First submitted 2011-01-02; First posted 2011-01-12 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: First Degree AV Block
Keywords: Implantable ICD; First Degree AV block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Device programming modifies AV timing (Experimental): DDD-40-BiV
  Interventions: Device: Cardiac resynchronization therapy-defibrillator
- Device programming allows intrinsic AV timing. (No Intervention): VVI-40-RV

INTERVENTIONS:
Device: Cardiac resynchronization therapy-defibrillator — Device programming that modifies AV timing
  Other Names: First degree AV block; Long PR interval
  Arms: Device programming modifies AV timing

SUMMARY:
The objective of the trial is to observe the effects of restoring atrioventricular (AV) synchrony in subjects with prolonged PR intervals. This will be assessed both acutely and chronically using echocardiographic and functional measurements.

DETAILED DESCRIPTION:
Same as above.

ELIGIBILITY:
Inclusion Criteria:

* Meet current indications for an implantable cardioverter-defibrillator (ICD) implant with:
* QRS width < 120 msec
* Left ventricular ejection fraction (LVEF) < 35% (no more than 180 days prior to enrollment)
* NYHA functional class II/III
* Optimal pharmacological heart failure therapy
* PR interval >/= 230 msec
* Ability to tolerate protocol required programming
* Access to a telephone line compatible with the LATITUDE® Communicator
* Subjects in sinus rhythm at the time of the baseline visit and who are expected to remain in sinus rhythm for the duration of the study
* Age 18 or above, or of legal age to give informed consent specific to state and national law
* Willing and capable of providing informed consent, undergoing a device implant, participating in all testing associated with this clinical investigation at an approved clinical investigational center and return to the investigational center at the intervals defined by this protocol

Exclusion Criteria:

* Previously placed pacemaker, ICD, or CRT device
* Inability or refusal to sign the Informed Consent Form
* Documented life expectancy of less than 12 months or expected to undergo heart transplant within the next 12 months
* Have tricuspid valve disease or who are likely to receive a mechanical tricuspid valve during the course of the clinical investigation
* Inability or refusal to comply with the follow-up schedule
* Have a neuromuscular, orthopedic, or other noncardiac condition that prevents subject from normal unsupported walking for the six minute hall walk test
* Have surgically uncorrected primary valvular heart disease
* Second or third degree atrioventricular block (AVB)
* Permanent or persistent atrial tachyarrhythmia that is refractory to all therapies
* Have had cardiac surgery, percutaneous coronary intervention, or myocardial infarction within 3 months of signing consent or who are likely to undergo a cardiac surgery or procedure in the foreseeable future
* Enrolled in any concurrent study unless written approval has been obtained from Boston Scientific or The Integra Group
* Women who are pregnant or plan to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Olshansky, MD, Principal Investigator — University of Iowa Hospitals; John Day, MD, Principal Investigator — Intermountain Medical Center

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Device Programming That Modifies AV Timing: Cardiac resynchronization therapy-defibrillator: Device programming that modifies AV timing
- Device Programming That Allows Intrinsic AV Timing.: Cardiac resynchronization therapy-defibrillator: Device programming that does not modifies AV timing
Period: Overall Study
Arm/Group | Device Programming That Modifies AV Timing | Device Programming That Allows Intrinsic AV Timing.
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Study terminated | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Device Programming Modifies AV Timing | Device Programming Allows Intrinsic AV Timing. | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Range Finding of Functional and Hemodynamic Changes Using Echocardiographic Determined Measures.
Description: Echocardiographic measures will include, but not be limited to, left ventricular volumes, left ventricular diameters, and ejection fraction.
Time Frame: 6 months
Population: The study was terminated early: long PR intervals are relatively rare in this population, and it would take an inordinately long time to enroll sufficient patients. Because of the early termination of the study, no data was analyzed since the primary objective is underpowered.
Arm/Group | Device Programming That Modifies AV Timing | Device Programming That Allows Intrinsic AV Timing.
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported as of ICF signature, and were supposed to be collected until the 12-month follow-up visit. However, the study was terminated early (1 subject had a 6-month follow-up visit, the second subject did not have a 6-month follw-up visit).
Description: An adverse event (AE) was defined as any undesirable clinical occurrence in a subject. This can be a subject complaint, change in health status, or product issue. An adverse event will not be reported if the underlying condition existed at enrollment and continued unchanged thereafter unless the event worsened considerably and required additional medical or pharmacological treatment.
Arm/Group | Device Programming That Modifies AV Timing | Device Programming That Allows Intrinsic AV Timing.
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device Programming That Modifies AV Timing (N=1) | Device Programming That Allows Intrinsic AV Timing. (N=1)
Sarcoidosis induced cardiomyopathy (Cardiac disorders) | 1 (2) | 0 (0)
Cataract surgery (Eye disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device Programming That Modifies AV Timing (N=1) | Device Programming That Allows Intrinsic AV Timing. (N=1)
Prolonged hospitalization due to sarcoidosis induced cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Dizziness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Non-sustained ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small number of patients analyzed. As the study was stopped early, the primary objective is underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No